CLINICAL TRIAL: NCT04651504
Title: Implementing Multilevel Colon Cancer Screening Interventions to Reduce Rural Cancer Disparities
Brief Title: Rural Colon Cancer Screening Toolkit Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: 202010206; 5R01CA233848-02 (NIH)
Record Dates: First submitted 2020-11-25; First posted 2020-12-03 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-10

CONDITIONS: Colon Cancer Screening

STUDY DESIGN:
Intervention Model Description: This is a stepped wedge trial where clusters of sites sequentially enter the intervention. Independent samples of patients are enrolled within a cluster at each set interval of time thus, it is analyzed as a repeated cross-sectional study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Primary Care Clinics (Experimental): * Southern Illinois Healthcare System will contact the site management and ask for participation in the study
  * Eligible providers and staff will be identified by clinic management. The research coordinator will work with the clinic to schedule a virtual site visit(s). The study team will interview providers and staff at the beginning and/or end of each active intervention period to assess knowledge and attitudes about CRC screening and follow-up processes, the Consolidated Framework for Implementation Research (CFIR) constructs such as role clarity within the clinical team, and satisfaction with the intervention and implementation. Post-implementation surveys will also ask about work-arounds and adaptations of the intervention tools and perceived efficacy.
  Interventions: Other: Colorectal Cancer Toolkit

INTERVENTIONS:
Other: Colorectal Cancer Toolkit — The intervention toolkit will include patient education materials and supportive materials for providers. Tracking systems and supports will be jointly developed with participating clinic and providers, in order to maximize their existing systems and develop processes that meet their needs and preferences, and training will be offered to help providers/teams efficiently use the tracking system and clinic resources. The study team will provide technical assistance and support through email, phone and zoom to support the clinic in their implementation process.

SUMMARY:
Less than half of all positive fecal immunochemical testing (FIT)s are followed-up by colonoscopy, thus limiting the full potential of colorectal cancer (CRC) screening to reduce mortality. Given the need for coordination in order to achieve high rates of follow-up, multilevel approaches are needed. Such approaches could be particularly beneficial in communities and populations that experience cancer disparities and have fewer specialty providers, but most data focuses on large systems or urban areas. The academic-community health system collaboration is uniquely poised to address this research and service gap. The persistent poverty and health disparities in rural Southern Illinois set the stage for truly impactful research. The investigators' approach will serve as a model for multilevel interventions in rural settings, inform future work addressing other health disparities, and fill a gap in rigorous trials of CRC screening follow-up in rural areas.

ELIGIBILITY:
Inclusion Criteria for Primary Care Clinic Sites

* Physician Hospital Organization (PHO) affiliated with Southern Illinois Healthcare

Exclusion Criteria for Primary Care Clinic Sites

* Not a part of the PHO

Inclusion Criteria for Physicians and Staff at Primary Care Clinic Sites

* Employment at the relevant clinic at the time of the study

Exclusion Criteria for Physicians and Staff at Primary Care Clinic Sites

* Not employed at the relevant clinic at the time of the study

Inclusion Criteria for Patients

* Age 45-75 during the study period
* Must be patient of the selected primary care clinic sites

Exclusion Criteria for Patients

* Younger than 45 years of age or older than 75 years of age during the study period
* Not a patient of the selected primary care clinic sites

Inclusion Criteria for Community Members

* Age 45-75 at the time of the health fair or screening event
* Able to undergo stool testing as determined by SIH staff at the health fair or screening event

Exclusion Criteria for Community Members

* Younger than 45 years of age or older than 75 years of age
* Unable to undergo stool testing

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 185903 (Actual)
Dates: Start 2020-12-02 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Number of referrals for colonoscopies after positive fecal immunochemical test | Completion of follow-up (estimated to be 44 months)
Number of colonoscopy completions after positive fecal immunochemical test | Completion of follow-up (estimated to be 44 months)
  -Within 60 days of referral

SECONDARY OUTCOMES:
Time to colonoscopy | Completion of follow-up (estimated to be 44 months)
Proportion of participants who initiate a colonoscopy within 14 days of positive fecal immunochemical test | Completion of follow-up (estimated to be 44 months)
Proportion of patients who complete a complete diagnostic evaluation within 60 days of positive fecal immunochemical test | Completion of follow-up (estimated to be 44 months)

CONTACTS AND LOCATIONS:
Overall Officials: Aimee James, Ph.D., MPH, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

DOCUMENTS (1):
  • Informed Consent Form (2020-11-25): https://cdn.clinicaltrials.gov/large-docs/04/NCT04651504/ICF_000.pdf